CLINICAL TRIAL: NCT06936592
Title: How Can Prefabricated Membrane-loaded Ascorbic Acid Curtail the Gingival Recession?
Brief Title: How Can Prefabricated Membranes Load Ascorbic Acid Can Curtail Gingival Recession?
Acronym: recession
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, shaimaa hamdy, lecturer of periodontology, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: gingival recession treatment; committe no 109 (Other: faculty of dentistry minia university)
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-01

CONDITIONS: Gingival Recession, Localized; Gingival Diseases; Recession, Gingival
Keywords: recession; membrane; ascorbic acide; graft
MeSH Terms: conditions — Gingival Recession; Gingival Diseases | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Inclusion criteria:
  1. Patients of both genders with ages more than 18 years.
  2. At least two adjacent teeth in maxillary or mandibular anterior sextant with Cairo classification (RT1 or RT 2) labial GR defect.
  3. Good general health with no contraindications for periodontal surgery (American Society of Anesthesiologists I).
  4. Non-smoker patients.
  Exclusion criteria:
  1. Pregnant and lactating women.
  2. Mal alignment teeth.
  3. Patients under active orthodontic therapy.
  4. Periodontal therapy during the last 6 months.
  Groups and intervention:
  Patients selected in this study will be classified into two groups:
  • Group 1: Fifteen patients will receive Phase I therapy; reevaluation after four weeks then will be treated with a placebo membrane
Who Masked: Participant, Outcomes Assessor
Masking Description: participants do not know the type of membrane and the outcomes assessor does not know type of group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Fifteen patients will receive Phase I therapy; reevaluation after four weeks then will be treated with a placebo membrane
  Interventions: Drug: Ascorbic acid
- study group (Active Comparator): Fifteen patients will receive Phase I therapy; reevaluation after four weeks then will be treated with membrane loaded by Ascorbic acid
  Interventions: Drug: Ascorbic acid

INTERVENTIONS:
Drug: Ascorbic acid — Ascorbic acid induce gingival healing

SUMMARY:
Periodontal diseases are a prevalent issue, often leading to gingival recession, where the gingival margin recedes, exposing the tooth root and causing various problems. Gingival recession can be managed through both non-surgical and surgical interventions The non-surgical approach often involves plaque control and addressing any underlying inflammatory conditions. However, in cases of advanced recession, surgical treatment may be necessary Several treatment techniques have been proposed, which can be divided into pedicle and free grafts. The latter can also be classified as free gingival grafts (FGG) or as connective tissue grafts (CTG). Other treatment options include soft tissue substitutes or regenerative therapies Harvesting graft from the palate has several problems, such as pain, inflammation, bleeding, flap necrosis, and infection at the donor site. For this reason, we need a substitute for soft tissue graft harvesting Carbopol polymers, also known as carbomers, are widely utilized in pharmaceutical formulations for their excellent mucoadhesive properties. This high molecular weight, cross-linked acrylic acid polymers are particularly effective in enhancing the adhesion of formulations to mucosal surfaces, thereby improving drug delivery and bioavailability

DETAILED DESCRIPTION:
Gingival recession is a common finding in daily clinical practice. Several issues may be associated with the apical shift of the gingival margin such as dentine hypersensitivity, root caries, non-carious cervical lesions (NCCLs), and compromised aesthetics. The first step in an effective management and prevention program is to identify susceptibility factors and modifiable conditions associated with gingival recession. Non-surgical treatment options for gingival recession defects include establishing optimal plaque control, removing overhanging subgingival restorations, behavior change interventions, and using desensitizing agents. In cases where a surgical approach is indicated, coronally advanced flap and tunneling procedures combined with a connective tissue graft are considered the most predictable treatment options for single and multiple recession defects. If there is a contraindication for harvesting a connective tissue graft from the palate or the patient wants to avoid a donor site surgery, adjunctive use of acellular dermal matrices, collagen matrices, and/or enamel matrix derivatives can be a valuable treatment alternative. For gingival recession defects associated with NCCLs a combined restorative-surgical approach can provide favourable clinical outcomes. If a patient refuses a surgical intervention or there are other contraindications for an invasive approach, gingival conditions should be maintained with preventive measures. This paper gives a concise review of when and how to treat gingival recession defects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders with ages more than 18 years.
2. At least two adjacent teeth in maxillary or mandibular anterior sextant with Cairo classification (RT1 or RT 2) labial GR defect.
3. Good general health with no contraindications for periodontal surgery (American Society of Anesthesiologists I).
4. Non-smoker patients.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Teeth exhibiting pathologic mobility.
3. Mal alignment teeth.
4. Patients under active orthodontic therapy.
5. Periodontal therapy during the last 6 months.
6. Patients received antibiotics or non-steroidal anti-inflammatory drugs six months before the beginning of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-17 (Estimated); Primary Completion 2025-10-17 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Gingival recession height | baseline, 3months and 6 months
  The distance from the cementoenamel junction to the gingival margin

IPD SHARING:
Plan to Share IPD: No
after study acceptance for journal all data about the study will be available

REFERENCES:
- [Background] Imber JC, Kasaj A. Treatment of Gingival Recession: When and How? Int Dent J. 2021 Jun;71(3):178-187. doi: 10.1111/idj.12617. Epub 2021 Jan 29. PMID 34024328
- See also: Treatment of Gingival Recession: When and How? — https://pmc.ncbi.nlm.nih.gov/articles/PMC9275303/